CLINICAL TRIAL: NCT03274193
Title: Effects of Yoga Training on Cardiovascular Reactivity to Psychological Stress in Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20170087
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (Experimental): The yoga group will engage in the yoga training program which is 60 minutes per session, 2 times per week for 12 weeks.
  Interventions: Behavioral: Yoga training program
- Control (No Intervention): The control group will be asked not to participate in any exercise program during the course of the study.

INTERVENTIONS:
Behavioral: Yoga training program — The hatha yoga program will be led by an experienced yoga instructor. Each 60 minutes session will consist of 10 minutes of breathing exercises (pranayama), 40 minutes of yoga pose practice (asana), and 10 minutes of supine meditation/relaxation (savasana). Yoga props, such as blocks and belts, will be used in accordance to each participant's particular body type and needs to help he/she achieve precise yoga postures safely and comfortably. The yoga poses are chosen for providing a restorative session and based on their purported relationship to restorative effects. Participants will be instructed to maintain their concentration and breath control at all times during the yoga session.
  Arms: Yoga

SUMMARY:
The purpose of this study is to examine the effects of 12-week yoga training on blood pressure, heart rate, heart rate variability, arterial stiffness, and total peripheral resistance during rest and psychological stress in patients with hypertension. All eligible participants will be randomly assigned to either yoga (n=40) or usual care control (n=40) group. During the 1st lab visit, the experimenter will explain the purpose and procedures of the study. If the participants understand and agree to participate in this study, they will be asked to sign the informed consent. Next, participants will fill out questionnaires, including demographic information, Physical Activity Readiness Questionnaire, perceived stress scale, anxiety inventory, exercise behavior questionnaire, and quality of life scale. Participant's resting blood pressure will be measured. Participants will then be instructed to relax in a supine position for 15 minutes while ECG is recording. Next, participants will perform 5 minutes of stroop task and 5 minutes of mental arithmetic task (mental stressors). ECG and cardiac output will be monitored throughout the whole session. After the stress period, participants will be asked to relax until heart rate becomes stable and return to baseline. The participants will perform the sit-and-reach test. After completing all the baseline testing, the yoga group will begin the training program which is 60 minutes per session, 2 times per week for 12 weeks. The control group will be asked not to participate in any exercise program during the course of the study. Participants will be filling out the same questionnaires and receive measures of blood pressure, ECG, and cardiac output at week 6 and week 12. Additionally, participants will perform the stress tasks and the sit-and-reach test again at week 12.

ELIGIBILITY:
Inclusion Criteria:

* 20-65 years of age
* 18.5 <=BMI<=29.9
* have hypertension (clinical diagnosis)
* resting systolic blood pressure 120-160 mmHg, resting diastolic blood pressure lower than 110 mmHg

Exclusion Criteria:

* regular exercise behaviors or current participation in yoga programs
* have cardiovascular diseases, pulmonary diseases, diabetes
* have musculoskeletal problems that may affect yoga pose practice (e.g., herniated intervertebral disc, spondylolithesis, ankylosing spondylitis)
* current pregnancy or breastfeeding
* change of hypertension medication use within 4 weeks

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure during rest from baseline to week 13 | Blood pressure during rest will be measured at baseline and week 13.
  Blood pressure will be assessed with an OMRON blood pressure monitor.

SECONDARY OUTCOMES:
Change in blood pressure during psychological stress from baseline to week 13 | Blood pressure during psychological stress will be measured at baseline and week 13.
  Blood pressure will be assessed with an OMRON blood pressure monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No